CLINICAL TRIAL: NCT03468868
Title: Comparative Effectiveness Study of an Exercise Intervention Delivered Via Telerehabilitation and Conventional Mode of Delivery
Brief Title: Comparative Effectiveness Study Telerehab Versus Conventional
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: University of Alabama at Birmingham (Other); University of North Carolina, Chapel Hill (Other); University of Georgia (Other); The Cleveland Clinic (Other); University of Colorado, Denver (Other); Marquette University (Other); Accelerated Cure Project for Multiple Sclerosis (Other); Patient-Centered Outcomes Research Institute (Other); Tanner Foundation for Multiple Sclerosis (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Deborah Backus, Director of Multiple Sclerosis Research, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS-1610-36999
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Exercise; Physical activity; Telerehabilitation; Comparative effectiveness study; Social cognitive theory; Health behavior change
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two-stage randomized choice design aimed at noninferiority.
Who Masked: Outcomes Assessor
Masking Description: Evaluators who assess clinical reported outcomes will be blinded to arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facility-based rehabilitation (Active Comparator): Participants will conduct the exercise program for people with MS in a facility, for example a gym, or rehabilitation center. They will receive coaching on site at the facility.
  Interventions: Behavioral: Exercise program for people with MS
- Telerehabilitation (Active Comparator): Participants will conduct the exercise program for people with MS at home and receive coaching via phone or Skype sessions.
  Interventions: Behavioral: Exercise program for people with MS

INTERVENTIONS:
Behavioral: Exercise program for people with MS — The intervention consists of 30 minutes of resistance training and 30 minutes of cardio three times per week for 16 weeks.

SUMMARY:
This study aims to compare the effectiveness of an exercise program delivered in a conventional facility-based format versus a telerehabilitation format, which takes place in the home. Exercise can improve mobility and perhaps decrease the rate and extent of disability in people with MS. Evidence shows that traditional, facility-based exercise training may help people with MS consistently participate in exercise or to exercise at a higher, more intense level. Despite this evidence, lack of access to facility-based exercise programs may make it difficult for people with MS to engage in exercise.Telerehabilitation (telerehab) has great potential to overcome challenges associated with facility-based programs. Telerehab can include videoconferencing, remote monitoring of signs and activity, and dissemination of specialized and individualized information via electronic mechanisms, such as smartphones and computers. Both facility-based and telerehab exercise training have yielded positive results in people with MS, but have not been compared head-to-head. The current study will fill this gap in the evidence base and compare the outcomes of delivering the same exercise interventions in a facility or in the home/community using a telerehab approach. The interventions are designed to be identical in content, with the only difference being the mode of training delivery.

DETAILED DESCRIPTION:
Funded by Patient-Centered Outcomes Research Institute (PCORI), this four-year, multi-site study aims to compare the effectiveness of a 16-week telerehabilitation (telerehab) exercise program and a facility-based exercise program on Multiple Sclerosis (MS) outcomes. The research study design is a two-stage randomized choice design aimed at non-inferiority.

Four hundred participants with MS who have ambulatory difficulties will be recruited from nine sites. First level randomization will assign participants to one of two groups - Choice or Random. The participants in Choice will be able to choose in which program they wish to participate (telerehab or facility-based). Individuals in the Random group, will be further randomized to either the telerehab or facility-based program. The research protocol and associated tools will be reviewed and approved by all relevant Research Review Committees before any research takes place. The study will comply with best practices in human subjects' research including following HIPAA guidelines and using strict informed consent procedures. Clinical reported outcome measures and patient reported outcome measures will be administered at baseline, immediately post-intervention (at 16 weeks), and at 12 months post-intervention. Patient reported outcomes will also be administered at 2 months and 6 months after the start of the intervention.

Dr. Deborah Backus is the principal investigator (PI) and Prof. Robert Motl is the co-Principal Investigator supported by collaborating co-Investigators at the Cleveland Clinic Mellen Center, Ohio; Marquette University, Wisconsin; University of Colorado, Denver; University of North Carolina, Chapel Hill; the University of Georgia; the Tanner Center for Multiple Sclerosis, Birmingham Alabama; Massachusetts General Hospital, Boston, Massachusetts; and the iConquerMS outcomes data collaborative (Accelerated Cure Project for MS). Shepherd Center is the primary and coordinating site for all study activities under Dr. Backus. University of Alabama at Birmingham (UAB) under the leadership of Prof. Motl will oversee delivery of the training programs, and statistical analysis under the direction of Dr. Gary Cutter.

This study will yield important data regarding the comparative impact of exercise programs on MS outcomes and provide information to people with MS, health providers, payers, exercise partners, and policy makers about how people with MS who have ambulatory difficulties can safely and effectively exercise.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate MS
* Has limitations in walking but can walk 25 feet
* Does not participate in a rigorous exercise program
* Can travel to trial site for assessments and training

Exclusion Criteria:

* Relapse in the past 30 days
* Other neurological or musculoskeletal disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Backus, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (9):
- United States (9):
  - The Tanner Center for Multiple Sclerosis, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - University of Colorado, Denver, Colorado
  - University of Georgia, Athens, Georgia
  - Shepherd Center, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Marquette University, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motl RW, Backus D, Neal WN, Cutter G, Palmer L, McBurney R, Schmidt H, Bethoux F, Hebert J, Ng A, McCully KK, Plummer P. Rationale and design of the STEP for MS Trial: Comparative effectiveness of Supervised versus Telerehabilitation Exercise Programs for Multiple Sclerosis. Contemp Clin Trials. 2019 Jun;81:110-122. doi: 10.1016/j.cct.2019.04.013. Epub 2019 Apr 22. PMID 31022481
- [Background] Neal WN, Moldavskiy M, Truax B, Ithurburn A, Ware M, Hebert JR, Opielinski L, Penko AL, Kern K, Palmer L, Backus D, Motl RW. Intervention fidelity and adaptation in a multi-site exercise training intervention for adults with multiple sclerosis. Contemp Clin Trials. 2023 Oct;133:107320. doi: 10.1016/j.cct.2023.107320. Epub 2023 Aug 24. PMID 37633458
- [Background] Palmer LC, Neal WN, Motl RW, Backus D. The Impact of COVID-19 Lockdown Restrictions on Exercise Behavior Among People With Multiple Sclerosis Enrolled in an Exercise Trial: Qualitative Interview Study. JMIR Rehabil Assist Technol. 2022 Nov 22;9(4):e42157. doi: 10.2196/42157. PMID 36269870
- [Background] Motl RW, Plummer P, Backus D, Hebert JR, Neal WN, Ng A, Lowman J, Bethoux F, Schmidt H, McBurney R, McCully KK, Cutter G. Validation of scores from a telephone administered multiple sclerosis walking scale-12 in persons with multiple sclerosis. Mult Scler Relat Disord. 2024 Aug;88:105715. doi: 10.1016/j.msard.2024.105715. Epub 2024 Jun 9. PMID 38889558
- [Derived] Motl RW, Backus D, Hebert JR, Ng AV, McCully KK, Neal WN, Schmidt H, McBurney R, Plummer P, Bethoux F, Lowman J, Cutter G. Walking performance is worse in black than white people with multiple sclerosis. Mult Scler Relat Disord. 2025 Mar;95:106343. doi: 10.1016/j.msard.2025.106343. Epub 2025 Feb 18. PMID 39986137
- [Derived] Motl R, Neal W, Backus D, Hebert J, McCully K, Bethoux F, Plummer P, Ng A, Lowman J, Schmidt H, McBurney R, Cutter G. Middle-range scores from the patient determined disease steps scale reflect varying levels of walking dysfunction in multiple sclerosis. BMC Neurol. 2024 Oct 10;24(1):383. doi: 10.1186/s12883-024-03871-1. PMID 39390466

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Started | 198 | 181
Completed | 151 | 115
Not Completed | 47 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Facility-based Rehabilitation | Telerehabilitation | Total
Number analyzed (Participants) | 198 | 181 | 379
Age, Categorical [Count of Participants; unit: Participants] — To qualify for this study, participants must have been aged 18 - 65.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 198 | 181 | 379
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — To qualify for this study, participants must have been aged 18 - 65.
  years | 51.47 (10.01) | 50.08 (9.18) | 50.81 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 value is missing in Gender.
  Participants
    number analyzed (Participants) | 198 | 180 | 378
    Female | 144 | 142 | 286
    Male | 54 | 38 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 185 | 170 | 355
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 50 | 105
  White | 126 | 120 | 246
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 10 | 6 | 16
MS type [Count of Participants; unit: Participants] — Population: 28 values are missing for MS type.
  Participants
    number analyzed (Participants) | 184 | 167 | 351
    Primary Progressive Multiple Sclerosis (PPMS) | 17 | 21 | 38
    Progressive Relapsing Multiple Sclerosis (PRMS) | 2 | 4 | 6
    Relapsing Remitting Multiple Sclerosis (RRMS) | 143 | 112 | 255
    Secondary Progressive Multiple Sclerosis (SPMS) | 22 | 30 | 52
Employment Status [Count of Participants; unit: Participants]
  Employed | 66 | 67 | 133
  Unemployed | 87 | 87 | 174
  Other | 45 | 27 | 72
Living Arrangement [Count of Participants; unit: Participants] — Population: 2 values are missing for Living Arrangement.
  Participants
    number analyzed (Participants) | 196 | 181 | 377
    Living Alone | 43 | 40 | 83
    Living With Others | 153 | 141 | 294
Patient-Determined Disease Steps (PDDS) Scale [Count of Participants; unit: Participants] — The Patient-Determined Disease Steps (PDDS) scale is a patient-reported measure of disability due to multiple sclerosis (MS). The scale focuses mainly on how well individuals with MS walk. Scores range from 0 (normal function) to 8 (bedridden). Higher scores reflect greater disability due to MS.
  Participants
    1 (Mild Disability) | 0 | 1 | 1
    3 (Gait Disability) | 55 | 48 | 103
    4 (Early Cane) | 67 | 57 | 124
    5 (Late Cane) | 45 | 49 | 94
    6 (Bilateral Support) | 31 | 26 | 57
Insurance [Count of Participants; unit: Participants]
  Direct purchase | 10 | 10 | 20
  Employer | 80 | 78 | 158
  Medicare | 59 | 52 | 111
  Medicaid | 29 | 31 | 60
  No insurance | 2 | 3 | 5
  Other | 18 | 7 | 25
Short Assessment of Health Literacy-English (SAHL-E) [Mean (Standard Deviation); unit: units on a scale] — The SAHL-E is an 18-item assessment of an English-speaking adult's ability to read and understand common medical terms. To be considered correct, the item must be pronounced correctly and accurately associated with a related term.
  Scores range from 0 (minimum) to 18 (maximum), with higher scores representing a greater ability to read and understand medical terms. A score between 0 and 14 suggests low health literacy.
  units on a scale | 17.51 (1.19) | 17.68 (0.61) | 17.59 (0.96)
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental Status Examination (MMSE) is a screening tool for cognitive impairment. Scores on the MMSE range from 0 (minimum) to 30 (maximum).
  Lower scores indicate greater cognitive impairment. Levels of impairment have been classified as (Tombaugh & McIntyre, 1992) as:
  Normal cognitive functioning: 24-30 Mild cognitive impairment: 18-24 Severe cognitive impairment: 0-17
  Participants were excluded from the study if their MMSE score was < 19.
  units on a scale | 29.33 (1.16) | 29.43 (0.99) | 29.38 (1.08)

OUTCOME MEASURES:

1. Primary Outcome: Timed 25 Foot Walk Test (T25FWT)
Description: The Timed 25 Foot Walk Test (T25FWT) is a measure of walking speed. Individuals are instructed to walk 25 feet as quickly and safely as possible from one marked end to the other.
  Higher walking speed (feet per second) indicate improved walking function.
Time Frame: Change from baseline T25FWT at 16-weeks
Population: Due to the COVID pandemic, some participants were unable or unwilling to return for in-person assessments following the intervention. Additionally, we noted differential attrition rates and participation in outcome assessments across the two groups.
Measure: Mean (Standard Deviation); unit: feet per second
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
feet per second
  Walking speed at baseline | 2.88 (0.85) | 2.62 (0.94)
  Walking speed at 16 weeks: number analyzed (Participants) | 137 | 92
  Walking speed at 16 weeks | 3.41 (1.12) | 3.26 (1.08)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Non-Inferiority — We chose a non-inferiority margin of 10% (or 0.10 feet per second) for this population; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.14 to 0.44], Standard Deviation 1.10

2. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The six minute walk test (6MWT) assesses walking endurance and aerobic capacity. The score is the distance walked in 6 minutes. Higher scores (more distance walked in feet) indicate improved walking capacity.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
feet
  Walking distance at baseline | 963.3 (381.1) | 884.2 (392.3)
  Walking distance at 16 weeks: number analyzed (Participants) | 137 | 92
  Walking distance at 16 weeks | 1099.6 (395.1) | 1027.1 (367.0)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = 72.46, 95% CI 2-sided [-29.56 to 174.5], Standard Deviation 384.1

3. Secondary Outcome: Multiple Sclerosis Walking Scale (MSWS)-12 Questionnaire
Description: The MSWS-12 is a self-reported measure of the impact of multiple sclerosis (MS) on walking ability and daily activities over the past two weeks. Items are scored from 1-5, with 1 meaning no limitation and 5 meaning extreme limitation.
  Scores are calculated by first adding the responses, and getting a total score of 12 - 60. This score is then transformed to a 0 - 100 scale (Nilsagard et al, 2007) by subtracting 12 from the sum, dividing by 48, and then multiplying by 100.
  Higher scores indicate a greater impact of MS on walking than lower scores.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 197 | 179
score on a scale
  MSWS at baseline | 61.36 (21.81) | 62.45 (22.35)
  MSWS at 16 weeks: number analyzed (Participants) | 150 | 113
  MSWS at 16 weeks | 53.54 (24.83) | 58.25 (25.14)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = -4.71, 95% CI 2-sided [-10.84 to 1.41], Standard Deviation 24.96

4. Secondary Outcome: Godin Leisure-Time Physical Activity (LTPA) Questionnaire
Description: The Godin LTPA is a 4-item, self-administered questionnaire assessing leisure-time physical activity. 3 questions ask how many times the individual participated in mild/light (e.g. yoga, easy walking), moderate (e.g. tennis, fast walking), and/or strenuous (e.g. running, basketball) activities in the past 7 days. The 4th question asks how often in a typical 7-day period the individual participates in an activity long enough to break a sweat (often, sometimes, or never/rarely).
  More strenuous activities are more heavily weighted. Total leisure activity score is calculated by multiplying the number of strenuous activities by 9, the number of moderate activities by 5, and the number of mild activities by 3, and then adding those scores together.
  A higher score means that the individual participates in more and/or more vigorous leisure-time physical activity. 24 units or more = active; 14-23 units = moderately active; < 14 units = sedentary.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
units on a scale
  LTPA at baseline | 7.48 (8.15) | 7.56 (8.01)
  LTPA at 16 weeks: number analyzed (Participants) | 151 | 115
  LTPA at 16 weeks | 23.09 (17.70) | 22.21 (18.88)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-3.55 to 5.32], Standard Deviation 18.22

5. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QOL) Survey
Description: Domains (anxiety, depression, fatigue, upper extremity function, lower extremity function, cognitive function, emotional and behavioral dyscontrol, sleep disturbance, ability to participate in social roles and activities, satisfaction with social roles and activities, stigma) - possible score of 8-40. Positive affect domain has possible score of 9-45. Communication domain has possible score of 5-25. No clinical thresholds established. Higher scores indicate WORSE self-reported health for Anxiety, Depression, Fatigue, Emotional and Behavioral Dyscontrol, Sleep Disturbance, Stigma. Higher scores indicate BETTER self-reported health for Upper Extremity Function, Lower Extremity Function, Cognitive Function, Positive Affect & Well-Being, Ability to Participate in Social Roles and Activities, Satisfaction with Social Roles & Activities, Communication.
Time Frame: Change from baseline at 16 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
units on a scale
  Baseline Anxiety Domain | 16.88 (7.01) | 17.19 (7.28)
  16 week Anxiety Domain: number analyzed (Participants) | 151 | 115
  16 week Anxiety Domain | 15.41 (6.86) | 14.75 (6.50)
  Baseline Depression Domain | 13.58 (6.14) | 13.90 (6.58)
  16 week Depression Domain: number analyzed (Participants) | 151 | 115
  16 week Depression Domain | 12.56 (6.20) | 12.31 (6.10)
  Baseline Fatigue Domain | 23.74 (7.58) | 24.96 (7.17)
  16 week Fatigue Domain: number analyzed (Participants) | 151 | 115
  16 week Fatigue Domain | 21.44 (7.85) | 22.31 (7.12)
  Baseline Upper Extremity Function Domain | 36.71 (4.09) | 36.78 (4.09)
  16 week Upper Extremity Function Domain: number analyzed (Participants) | 151 | 115
  16 week Upper Extremity Function Domain | 37.12 (4.08) | 37.06 (3.49)
  Baseline Lower Extremity Function Domain | 30.53 (5.26) | 30.17 (5.21)
  16 week Lower Extremity Function Domain: number analyzed (Participants) | 151 | 115
  16 week Lower Extremity Function Domain | 33.04 (5.22) | 31.52 (5.72)
  Baseline Cognitive Function Domain | 30.46 (7.55) | 30.41 (7.09)
  16 week Cognitive Function Domain: number analyzed (Participants) | 151 | 115
  16 week Cognitive Function Domain | 31.35 (7.52) | 32.24 (6.14)
  Baseline Emotional and Behavioral Dyscontrol Domain | 14.85 (5.84) | 14.66 (5.65)
  16 week Emotional and Behavioral Dyscontrol Domain: number analyzed (Participants) | 151 | 115
  16 week Emotional and Behavioral Dyscontrol Domain | 14.27 (6.14) | 13.19 (4.92)
  Baseline Positive Affect and Well-Being Domain | 35.20 (7.44) | 34.65 (7.14)
  16 week Positive Affect and Well-Being Domain: number analyzed (Participants) | 151 | 115
  16 week Positive Affect and Well-Being Domain | 36.55 (7.21) | 36.01 (7.03)
  Baseline Sleep Distrubance Domain | 18.29 (5.50) | 19.33 (6.11)
  16 week Sleep Distrubance Domain: number analyzed (Participants) | 151 | 115
  16 week Sleep Distrubance Domain | 16.76 (5.88) | 17.35 (5.61)
  Baseline Ability to Participate in Social Roles and Activities Domain | 29.44 (6.51) | 28.60 (7.04)
  16 week Ability to Participate in Social Roles and Activities Domain: number analyzed (Participants) | 151 | 115
  16 week Ability to Participate in Social Roles and Activities Domain | 30.77 (6.78) | 30.37 (6.48)
  Baseline Satisfaction with Social Roles and Activities Domain | 24.69 (7.85) | 24.57 (7.37)
  16 week Satisfaction with Social Roles and Activities Domain: number analyzed (Participants) | 151 | 115
  16 week Satisfaction with Social Roles and Activities Domain | 28.02 (7.60) | 27.37 (7.23)
  Baseline Stigma Domain | 15.28 (6.34) | 15.31 (5.75)
  16 week Stigma Domain: number analyzed (Participants) | 151 | 115
  16 week Stigma Domain | 13.74 (5.94) | 13.68 (5.31)
  Baseline Communication Domain | 21.88 (3.91) | 21.76 (3.89)
  16 week Communication Domain: number analyzed (Participants) | 151 | 115
  16 week Communication Domain | 22.07 (3.58) | 22.54 (3.26)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Anxiety Domain; Test type: Superiority; p = 0.43, t-test, 2 sided; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.97 to 2.30], Standard Deviation 6.71
Statistical Analysis 2: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Depression Domain; Test type: Superiority; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-1.26 to 1.74], Standard Deviation 6.16
Statistical Analysis 3: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Fatigue Domain; Test type: Superiority; p = 0.35, t-test, 2 sided; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-2.71 to 0.97], Standard Deviation 7.54
Statistical Analysis 4: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Upper Extremity Function Domain; Test type: Superiority; p = 0.91, t-test, 2 sided; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.88 to 0.99], Standard Deviation 3.83
Statistical Analysis 5: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Lower Extremity Function Domain; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [0.20 to 2.85], Standard Deviation 5.44
Statistical Analysis 6: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Cognitive Function Domain; Test type: Superiority; p = 0.29, t-test, 2 sided; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-2.54 to 0.76]
Statistical Analysis 7: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Emotional and Behavioral Dyscontrol Domain; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [-0.26 to 2.42]
Statistical Analysis 8: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Positive Affect and Well-Being Domain; Test type: Superiority; p = 0.54, t-test, 2 sided; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-1.19 to 2.28], Standard Deviation 7.13
Statistical Analysis 9: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Sleep Disturbance Domain; Test type: Superiority; p = 0.41, t-test, 2 sided; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-2.00 to 0.81], Standard Deviation 5.76
Statistical Analysis 10: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Ability to Participate in Social Roles and Activities Domain; Test type: Superiority; p = 0.63, t-test, 2 sided; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.22 to 2.02], Standard Deviation 6.65
Statistical Analysis 11: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Satisfaction with Social Roles and Activities Domain; Test type: Superiority; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-1.16 to 2.47], Standard Deviation 7.44
Statistical Analysis 12: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Stigma Domain; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.32 to 1.45], Standard Deviation 5.68
Statistical Analysis 13: Comparison: Facility-based Rehabilitation vs Telerehabilitation; NeuroQOL Communication Domain; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.31 to 0.37], Standard Deviation 3.45

6. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS)-29
Description: The MSIS measures individual's views on the impact of MS on day-to-day life during the past two weeks. It is comprised of two subscales: a 20-item physical impact scale and a 9-item psychological impact scale. The MSIS has no combined total score. Scores on the physical impact scale can range from 20 to 80 and on the psychological impact scale from 9 to 36.
  Lower scores indicate little impact of MS, and higher scores indicate a higher impact of MS (on either physical or psychological functioning).
Time Frame: Change from baseline at 16 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
units on a scale
  Baseline MSIS-29 Physical Scale | 39.63 (19.62) | 41.59 (18.24)
  16 week MSIS-29 Physical Scale: number analyzed (Participants) | 150 | 112
  16 week MSIS-29 Physical Scale | 32.18 (21.36) | 34.65 (19.61)
  Baseline MSIS-29 Psychological Scale | 31.71 (21.33) | 33.01 (22.16)
  16 week MSIS-29 Psychological Scale: number analyzed (Participants) | 150 | 112
  16 week MSIS-29 Psychological Scale | 24.79 (22.29) | 26.17 (20.06)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MSIS Physical; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-7.55 to 2.60], Standard Deviation 20.63
Statistical Analysis 2: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MSIS Psychological; Test type: Superiority; p = 0.24, t-test, 2 sided; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-6.63 to 3.88], Standard Deviation 21.37

7. Secondary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: The MFIS is a 21-item questionnaire that measures the impact of fatigue on the participant's activities and lifestyle over the past four weeks. Items on the MFIS can be broken into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. The physical subscale score can range from 0 to 36. The cognitive subscale score can range from 0 to 40. The psychosocial subscale score can range from 0 to 8. The total MFIS score is the sum total of all three subscales, and can range from 0 to 84.
  Higher scores indicate a greater impact of fatigue on a person's activities.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
score on a scale
  MFIS Cognitive at baseline | 14.54 (9.58) | 14.96 (9.06)
  MFIS Cognitive at 16 weeks: number analyzed (Participants) | 150 | 112
  MFIS Cognitive at 16 weeks | 12.00 (9.30) | 11.63 (8.36)
  MFIS Physical at baseline | 20.02 (7.81) | 20.98 (7.40)
  MFIS Physical at 16 weeks: number analyzed (Participants) | 150 | 112
  MFIS Physical at 16 weeks | 15.57 (8.21) | 17.67 (7.77)
  MFIS Psychosocial at baseline | 3.89 (2.20) | 3.97 (2.20)
  MFIS Psychosocial at 16 weeks: number analyzed (Participants) | 150 | 112
  MFIS Psychosocial at 16 weeks | 2.93 (2.20) | 3.07 (2.14)
  MFIS Total at baseline | 38.45 (17.36) | 39.91 (16.50)
  MFIS Total at 16 weeks: number analyzed (Participants) | 150 | 112
  MFIS Total at 16 weeks | 30.50 (18.02) | 32.37 (15.52)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MFIS Cognitive; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-1.83 to 2.56], Standard Deviation 8.91
Statistical Analysis 2: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MFIS Physical; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-4.07 to -0.12], Standard Deviation 8.03
Statistical Analysis 3: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MFIS Psychosocial; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.68 to 0.39], Standard Deviation 2.17
Statistical Analysis 4: Comparison: Facility-based Rehabilitation vs Telerehabilitation; MFIS Total; Test type: Superiority; p = 0.38, t-test, 2 sided; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-6.05 to 2.30], Standard Deviation 17.00

8. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. It characterizes disability level and determines disability progression in people with MS. Higher scores reflect greater disability due to MS.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
score on a scale
  EDSS at baseline | 5.32 (0.95) | 5.25 (0.94)
  EDSS at 16 weeks: number analyzed (Participants) | 137 | 92
  EDSS at 16 weeks | 5.02 (1.20) | 5.04 (1.16)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Superiority; p = 0.87, t-test, 2 sided; Mean Difference (Final Values) = -.03, 95% CI 2-sided [-0.34 to 0.29], Standard Deviation 1.18

9. Secondary Outcome: Patient Determined Disease Steps (PDDS)
Description: The PDDS is a patient-reported outcome of disability in MS. The scale focuses mainly on how well individuals with MS walk. Scores range from 0 (normal function) to 8 (bedridden). Higher scores reflect greater disability due to MS.
Time Frame: Change from baseline at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
Number analyzed (Participants) | 198 | 181
score on a scale
  PDDS at baseline | 4.26 (1.03) | 4.28 (1.04)
  PDDS at 16 weeks: number analyzed (Participants) | 151 | 115
  PDDS at 16 weeks | 1.66 (2.14) | 2.19 (2.31)
Statistical Analysis 1: Comparison: Facility-based Rehabilitation vs Telerehabilitation; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.08 to 0.00], Standard Deviation 2.21

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through the end of the 16 week intervention phase.
Description: During coaching sessions, the exercise coaches queried participants about any adverse events they experienced since the previous session. The site PI, study project manager, and study PI were notified of all AEs as they were reported.
Arm/Group | Facility-based Rehabilitation | Telerehabilitation
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/181
Serious Adverse Events (participants affected / at risk) | 8/198 | 2/181
Other Adverse Events (participants affected / at risk) | 80/198 | 88/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Facility-based Rehabilitation (N=198) | Telerehabilitation (N=181)
Coronavirus infections (Infections and infestations) | 2 (3) | 1 (1) — This SAE was determined to be not related to the study intervention.
Elective hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) — This SAE was determined to be not related to the study intervention.
Fall resulting in fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — This SAE was determined to be not related to the study intervention.
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — This SAE was determined to be not related to the study intervention.
Increase in multiple sclerosis (MS) symptoms (Nervous system disorders) | 1 (1) | 0 (0) — Participant missed an infusion of their disease-modifying therapy (DMT) which led to a severe increase in MS symptoms and hospitalization. This SAE was determined to be not related to the study intervention.
Septic shock of unknown etiology (Infections and infestations) | 1 (1) | 0 (0) — This SAE was determined to be not related to the study intervention.
Viral infection (Infections and infestations) | 1 (1) | 0 (0) — This SAE was determined to be not related to the study intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Facility-based Rehabilitation (N=198) | Telerehabilitation (N=181)
Coronavirus infection (Infections and infestations) | 8 (9) | 7 (8) — All were determined to be not related to the study intervention.
Dental conditions (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Reported conditions included pain (2) and a fractured tooth (1). All were determined to be not related to the study intervention.
Depression (Psychiatric disorders) | 0 (0) | 2 (2) — All were determined to be not related to the study intervention.
Fall with injury (Musculoskeletal and connective tissue disorders) | 25 (27) | 26 (32) — Injuries included minor skin abrasions, bruising, soreness, pain, sprain, fracture (3), and concussion (1). Of the 59 fall with injury events, 2 were determined to be possibly related, and 3 were determined to be related to the study intervention.
Fall without injury (General disorders) | 19 (22) | 16 (22) — Of the 44 fall without injury events, 3 were determined to be possibly related, and 8 were determined to be related to the study intervention.
Fatigue (Nervous system disorders) | 0 (0) | 4 (4) — Of the 4 fatigue events, 1 was determined to be possibly related, and 1 was determined to be related to the study intervention.
Gastroenteritis (Gastrointestinal disorders) | 4 (5) | 2 (2) — All were determined to be not related to the study intervention.
General illness (General disorders) | 1 (1) | 3 (3) — General illness included general, undiagnosed reports of feeling "sick". All were determined to be not related to the study intervention.
Heat intolerance (Nervous system disorders) | 1 (1) | 2 (2) — Of the 3 heat intolerance events, 1 was determined to be possibly related, and 1 was determined to be related to the study intervention.
Influenza Infection (Infections and infestations) | 1 (1) | 2 (2) — All were determined to be not related to the study intervention.
Medication side effects (Nervous system disorders) | 1 (1) | 3 (3) — All were determined to be not related to the study intervention.
Migraine (Nervous system disorders) | 0 (0) | 2 (2) — Of the 2 migraine events, 1 was determined to be possibly related to the study intervention.
Motor Vehicle Accident (MVA) with Sequelae (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — All were determined to be not related to the study intervention.
Multiple Sclerosis (MS) Flare (Nervous system disorders) | 2 (3) | 5 (5) — Of the 8 MS flare events, 1 was determined to be possibly related to the study intervention.
Multiple Sclerosis (MS) Relapse (Nervous system disorders) | 0 (0) | 2 (2) — Events were categorized as MS relapses only if diagnosed by a neurologist as such. All were determined to be not related to the study intervention.
Neurological Symptoms (Nervous system disorders) | 6 (6) | 2 (2) — Events included numbness (1), neuralgia (1), blurred vision (1), optic neuritis (1), increased spasticity (2), and worsening balance (2). Of the 8 neurological events, 5 were determined to be possibly related.
Other Musculoskeletal Conditions (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) — Events included swelling, tendonitis, sprain, and spinal stenosis. Of the 8 events, 3 were determined to be possibly related, and 1 was determined to be related to the study intervention.
Pain (Musculoskeletal and connective tissue disorders) | 19 (22) | 24 (26) — Pain was reported at the ankle (1), back (14), chest (3), elbow (1), foot (2), hip (3), knee (10), leg (2), neck (2), pelvis (1), shoulder (5), and thigh (1). Of the 48 events, 18 were possibly related, and 5 were related to the study intervention.
Symptoms post-COVID vaccine (Immune system disorders) | 3 (3) | 4 (5) — All were determined to be not related to the study intervention.
Upper respiratory infection (Infections and infestations) | 0 (0) | 9 (9) — All were determined to be not related to the study intervention.
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) — All were determined to be not related to the study intervention.
Vertigo (Nervous system disorders) | 2 (2) | 1 (1) — All were determined to be not related to the study intervention.
Weakness (Nervous system disorders) | 1 (1) | 5 (5) — Of the 6 reports of weakness, 5 were determined to be possibly related to the study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT03468868/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03468868/SAP_001.pdf